CLINICAL TRIAL: NCT06874465
Title: TAVI Registry at the National Research Center for Cardiac Surgery, Astana, Kazakhstan
Brief Title: Transcatheter Aortic Valve Implantation Registry at the National Research Center for Cardiac Surgery, Nur-Sultan, Kazakhstan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Cardiac Surgery, Kazakhstan (Other)
Collaborators: Medtronic Cardiovascular (Industry)
Responsible Party: Principal Investigator, Abdurashid, Head of the department of the catheterization laboratory, National Research Center for Cardiac Surgery, Kazakhstan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: v. 1; ERP-2019-11795 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2020-10-12; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients after transcatheter aortic valve replacement (Experimental): Patients after transcatheter aortic valve replacement
  We will compare TAVI with SAVR data on mortality, intraoperative complications, post-operative complications and adverse cardiovascular events. We will perform Quality of Life analysis before TAVI and one year later, using the Short-Form 36 (SF36) instrument on 70% of our patients.
  Interventions: Device: Transcatheter aortic valve implantation
- Patients after surgical aortic valve replacement (Active Comparator): Patients after surgical aortic valve replacement
  We will compare TAVI with SAVR data on mortality, intraoperative complications, post-operative complications and adverse cardiovascular events. We will perform Quality of Life analysis before TAVI and one year later, using the Short-Form 36 (SF36) instrument on 70% of our patients.
  Interventions: Device: Transcatheter aortic valve implantation

INTERVENTIONS:
Device: Transcatheter aortic valve implantation — Compare self expendable and balloon expendable valves
  Other Names: Surgical aortic valve replacement

SUMMARY:
This study will analyze patients with aortic stenosis who have undergone transcatheter valve implantation and surgical aortic valve replacement. Afterwards, the results of these two procedures will be collected to the database and compared among the Kazakhstani population.

DETAILED DESCRIPTION:
Primary Objectives

1. Prevalence of aortic stenosis in Kazakhstan regions
2. 12 months survival of patients after TAVI
3. Intra- and postoperative complications
4. Conduction disorders after TAVI
5. Left ventricle function after TAVI in patients with low ejection fraction
6. Comparison of aortic route dimensions by 3D-TEE and MSCT
7. Comparison of TAVR with SAVR

Study Design Registry, IV phase

Subject Follow-up Schedule Maximum follow-up is approximately 4 years.

Inclusion Criteria Patients have TAVI

Exclusion Criteria Patients have not TAVI

Primary Endpoints The database contains data on mortality, intraoperative complications, post-operative complications and adverse cardiovascular events. We will perform Quality of Life analysis before TAVI and one year later, using the Short-Form 36 (SF36) instrument on 70% of our patients.

Patient Safety The NRCCS is a leading center for interventional cardiology in Kazakhstan, and in Central Asia, performing a high volume of TAVI procedures annually

Procedure / Intervention Description

* We believe our database is unique because it is the first systematically-collected, prospectively designed database in Central Asia for patients receiving TAVI.
* As known there is no data has been published regarding TAVI in Central Asia.

Secondary Endpoints

* Surgeons at NRCCS tend to use biological valves over mechanical valves because it was recognized that the requirements for long term success of mechanical valves (e.g. warfarin maintenance and compliance) were unlikely to be achieved in our patient population, many of whom live in rural areas without access to advanced cardiology care.
* Some of these patients are now returning to our center for valve in valve implantation and are being included in our registry. • Foundational work has been completed through our database development, but there is significant potential to expand our data collection to other Central Asian interventional cardiology centers.
* As technology evolves and options for trans-femoral TAVI approaches increase, the likelihood of using TAVI over SAVR will increase in Kazakhstan and Central Asia.

Statistical Method / Rationale Foundational work has been completed through our database development, but there is significant potential to expand our data collection to other Central Asian interventional cardiology centers. As technology evolves and options for trans-femoral TAVI approaches increase, the likelihood of using TAVI over SAVR will increase in Kazakhstan and Central Asia.

ELIGIBILITY:
Inclusion Criteria:

* Patients has given written informed Concent for study participation prior to procedure
* Patients with Aortic Valve stenosis
* Patients has severe degenerative or congenital aortic stenosis.
* Patients has symptomatic aortic stenosis as demonstrated by NYHA II or greater

Exclusion Criteria:

* Patients has active endocarditis
* Patients has history of cerebral vascular accident or transient ischemic attack within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Number of death | 1 year
  12 month all-cause of mortality
Evaluate of echocardiographic results | 1 year
  echocardiographic parameters: Aortic valve orifice area, aortic valve bioprosthetic gradient (peak, mean), aortic valve bioprosthetic velocity, ejection fracrion of left ventricle (LVEF%).
Incidence of stroke | within 30 days and 12 months
  procedure associated stroke and 12 months
Permanent pacemaker implantation | within 30 days
  procedure associated AB block which is need for permanent pacemaker implantation

SECONDARY OUTCOMES:
Life quality | Baseline, 12 months
  Quality of life on 36-item short-form (SF 36) will be carry before and 12 months after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center for Cardiac Surgery, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No